CLINICAL TRIAL: NCT06460675
Title: Comparative Effects of Autogenic Inhibition and Reciprocal Inhibition Muscle Energy Techniques in Piriformis Syndrome
Brief Title: Comparasion of Autogenic Inhibition and Reciprocal Inhibition Muscle Energy Techniques (METS) in Piriformis Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/01114
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Piriformis Syndrome
Keywords: Exercise; Manipulative therapies; Pain; Piriformis Syndrome; Range of Motion; Sciatic Nerve
MeSH Terms: conditions — Piriformis Muscle Syndrome; Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenic Inhibition Muscle Energy Technique (Experimental): This group will receive Autogenic Inhibition Muscle Energy Technique
  Interventions: Procedure: Autogenic Inhibition Muscle Energy Technique; Procedure: Reciprocal Inhibition Muscle Energy Technique
- Reciprocal Inhibition Muscle Energy Technique (Active Comparator): This group will receive Reciprocal Inhibition Muscle Energy Technique
  Interventions: Procedure: Autogenic Inhibition Muscle Energy Technique; Procedure: Reciprocal Inhibition Muscle Energy Technique

INTERVENTIONS:
Procedure: Autogenic Inhibition Muscle Energy Technique — No of repetitions: 1 set with 3 repetitions No of Sessions per week: 2 per weeks for 3 weeks (40 Min per Session)
Procedure: Reciprocal Inhibition Muscle Energy Technique — No of repetitions: 1 set with 3 repetitions No of Sessions per week: 2 per week for 3 weeks (40 Min per Session)

SUMMARY:
To compare the effects of Autogenic Inhibition and Reciprocal Inhibition Muscle Energy Techniques (METS) in Piriformis Syndrome

DETAILED DESCRIPTION:
Piriformis syndrome is when the piriformis muscle, located in the buttock region, spasms and causes buttock pain. The piriformis muscle also can irritate the nearby sciatic nerve and cause pain, numbness, and tingling along the back of the leg and into the foot (similar to sciatic pain). The functional limitations experienced by hip pain patients in the lower limb profoundly impact their quality of life. This study aims to investigate the effectiveness of an integrated approach that compares the Effects of Autogenic Inhibition versus Reciprocal Inhibition Muscle Energy Techniques on Pain, Range of motion, and Disability in patients with Piriformis Syndrome.

This randomized clinical trial will be conducted at DHQ Hospital Jhang over six months. The sample size will consist of 32 participants. Participants who meet the inclusion criteria will be taken through a non-probability convenience sampling technique, that will be randomized through a sealed envelope method. 16 Participants will be assigned to Group A that will be treated with the Autogenic Inhibition Muscle Energy Technique, 16 Participants will be assigned to Group B and will be treated with Reciprocal Inhibition Muscle Energy Technique at the frequency of 1 set and 3 repetitions per session for two sessions per week and total six sessions for three weeks with follow up at one month. The duration of contraction is 7-10 seconds. Pre and post-intervention values will be taken on the 1st day in the 3rd week and at one-month follow-up. Data will be collected using various assessment tools, including the FAIR test, Freiberg test, Lasegue test, Beatty test, Pace sign, Numeric Pain Rating Scale (NPRS), and Universal Goniometer. Pre-intervention assessments will be conducted for all two groups. The effects of the interventions will be measured either by parametric or non-parametric tests after assessing the normality of data by the Shapiro-Wilk test Independent t-test. Data analysis will be performed by using SPSS 25 software.

ELIGIBILITY:
Inclusion Criteria:

* Both genders with ages between 25-45 years.
* Patients diagnosed with Piriformis syndrome using the Piriformis FAIR test, Freiberg test, Lasegue test, Beaty test, and pace sign.
* Hip pain with a threshold of NPRS 3-6.
* Limited ROM of Hip Internal Rotation and Abduction measured using a goniometer.
* Buttock pain ≥ 3 months.
* Pain with prolonged sitting (more than 20 minutes)

Exclusion Criteria:

* Hip Degenerative changes.
* History of Trauma or Fracture
* Other Systemic Conditions
* Postural abnormality/deformity
* Diagnosed Psychological Disorders
* Pregnancy

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-10 (Estimated); Study Completion 2024-11-10 (Estimated)

PRIMARY OUTCOMES:
Pain : Numeric Pain Rating Scale (NPRS) | 3 Weeks
  Patients' overall assessment of pain will be provided using the numeric pain rating scale
Range of Motion : Universal Goniometer | 3 Weeks
  It is frequently employed as a benchmark technique for the assessment of Range of Motion
Lower Extremity Functional Scale (LEFS) | 3 Weeks
  The LEFS is a self-report questionnaire intended to assess functional status in patients with disability of the lower extremity (e.g., hip, thigh, ankle) containing 20 questions about a person's ability to perform everyday tasks

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PhD, Principal Investigator — Riphah International University
Locations (1):
- IIMCT Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sadiq M, Hussain SA, Meganath P. 'Hand on hip'sign: A novel screening test and diagnostic tool in piriformis syndrome. Journal of Orthopaedics, Trauma and Rehabilitation. 2020:2210491720961113.
- [Background] Siahaan YMT, Tiffani P, Tanasia A. Ultrasound-Guided Measurement of Piriformis Muscle Thickness to Diagnose Piriformis Syndrome. Front Neurol. 2021 Sep 7;12:721966. doi: 10.3389/fneur.2021.721966. eCollection 2021. PMID 34557150
- [Background] Tanveer F, Shahid S. Frequency of Piriformis tightness in professionals middle aged women. Rawal Medical Journal. 2018;43(4):685-.
- [Background] Hopayian K, Danielyan A. Four symptoms define the piriformis syndrome: an updated systematic review of its clinical features. Eur J Orthop Surg Traumatol. 2018 Feb;28(2):155-164. doi: 10.1007/s00590-017-2031-8. Epub 2017 Aug 23. PMID 28836092
- [Background] Siahaan YMT, Ketaren RJ, Hartoyo V, Tiffani P. The predisposing factors of piriformis syndrome: Study in a referral hospital. MNJ (Malang Neurology Journal). 2019;5(2):76-9.
- [Background] Wu YY, Guo XY, Chen K, He FD, Quan JR. Feasibility and Reliability of an Ultrasound Examination to Diagnose Piriformis Syndrome. World Neurosurg. 2020 Feb;134:e1085-e1092. doi: 10.1016/j.wneu.2019.11.098. Epub 2019 Nov 25. PMID 31778837
- [Background] Islam F, Mansha H, Gulzar K, Raza A, Raffique A, Haider S. Prevalence Of Piriformis Muscle Syndrome Among Individuals with Low Back Pain: Piriformis Muscle Syndrome Among Individuals with Low Back Pain. Pakistan Journal of Health Sciences. 2022:48-52.
- [Background] Probst D, Stout A, Hunt D. Piriformis Syndrome: A Narrative Review of the Anatomy, Diagnosis, and Treatment. PM R. 2019 Aug;11 Suppl 1:S54-S63. doi: 10.1002/pmrj.12189. Epub 2019 Jul 22. PMID 31102324
- [Background] Ahmad Siraj S, Dadgal R. Physiotherapy for Piriformis Syndrome Using Sciatic Nerve Mobilization and Piriformis Release. Cureus. 2022 Dec 26;14(12):e32952. doi: 10.7759/cureus.32952. eCollection 2022 Dec. PMID 36712711
- [Background] Chang C, Jeno SH, Varacallo MA. Anatomy, Bony Pelvis and Lower Limb: Piriformis Muscle. 2023 Nov 13. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519497/ PMID 30137781